CLINICAL TRIAL: NCT04239430
Title: Evaluation of the Immunogenicity of Meningococcal B (4CMenB) and Meningococcal ACWY (MenACWY Conjugate) Vaccination in a Population With HIV at 18 and 30 Months After Two Doses of Vaccine
Brief Title: Propositive (Protecting Positive People From Meningococcal Infection) Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019.0374
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2021-07

CONDITIONS: HIV/AIDS; Meningococcal Disease
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Meningococcal Infections | interventions — Serum Bactericidal Antibody Assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum Bactericidal Assays — Blood samples will be taken from participants at two time points in the study. Serum Bactericidal Assays from participant serum using relevant MenB and MenACWY strains will be undertaken at 18 and 30 months post two doses of 4CMenB (Bexsero, GSK) and MenACWY-conjugate (Menveo, GSK) vaccine. The Vaccines were given to participants during an earlier clinical trial (Propositive). This trisal is a follow up study.

SUMMARY:
The need for and timing of booster doses of meningococcal vaccines in People Living with HIV (PLWHIV) is currently unknown. As such it is impossible for clinicians to recommend booster doses or to know if and when these might be necessary.We propose to follow up a group of participants from the Propositive study who received two doses of both MenB (Bexsero) and MenACWY (Menveo). This was a group of PLWHIV between the ages 18-45 years. We propose following up these participants at 18 and 30 months post completion of two doses of vaccine and investigating their immunological response.

ELIGIBILITY:
Inclusion Criteria:

* Received vaccination with Bexsero and Menveo during Propositive study
* Able to sign fully informed consent
* Able to comply with study requirements

Exclusion Criteria:

• Unwilling or unable to comply with study requirements

Ages: 18 Years to 47 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is the same as for the original Propositive study. This study will follow up the same cohort of participants.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Serum bacteridical Assay responses against relevant MenB strains at 18 and 30 months post two doses Bexsero (administered concomitantly with Menveo) | The 18 month blood test is taken 548 days (+/-60 days) from completion of vaccination during the Propositive study and the 30 month blood test is taken 912 days (+/- 60 days) after completion of vaccination
  1. Geometric Mean Titres against relevant MenB strains at 18 and 30 months post two doses of Bexsero
  2. The proportion of subjects with at least 4 fold increase in hSBA against relevant MenB strains from baseline compared to 18 month and 30 months post two doses of Bexsero
  3. The proportion of subjects with "protective" hSBA titres >4 against relevant MenB strains at 18 months and 30 months post two doses of Bexsero

SECONDARY OUTCOMES:
Serum bactericidal Assay responses against relevant MenACWY strains at 18 and 30 months post two doses Menveo (administered concomitantly with Bexsero) | The 18 month blood test is taken 548 days (+/-60 days) from completion of vaccination during the Propositive study and the 30 month blood test is taken 912 days (+/- 60 days) after completion of vaccination
  4. rSBA GMTs for MenACWY antigens at 18 and 30 months.
  5. The proportion of subjects with at least 4 fold increase in rSBA against relevant MenACWY serogroups from baseline compared to at 18 and 30 months.
  6. The proportion of subjects with "protective" rSBA titres >8 against relevant MenACWY serogroups at 18 and 30 months.

CONTACTS AND LOCATIONS:
Locations (1):
- St George's University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No